CLINICAL TRIAL: NCT05694312
Title: Ibrutinib for the Treatment of Autoimmune Hemolytic Anemia in Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma or CLL-like Monoclonal B-cell Lymphocytosis
Brief Title: Ibrutinib for the Treatment of AIHA in Patients With CLL/SLL or CLL-like MBL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL2323
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Autoimmune Hemolytic Anemia; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Monoclonal B-Cell Lymphocytosis CLL-Type
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ibrutinib (Experimental): Patients will receive ibrutinib 420 mg/day orally for up to 12 cycles of 28 days.
  Interventions: Drug: Ibrutinib 420 mg

INTERVENTIONS:
Drug: Ibrutinib 420 mg — Patients will receive ibrutinib orally on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of CLL progression or unacceptable toxicity.

SUMMARY:
This is a multicenter, single arm, phase II study aimed at evaluating ibrutinib therapy for the treatment of AIHA in patients with CLL/SLL or CLL-like MBL.

DETAILED DESCRIPTION:
This is a multicenter, phase II study to assess the efficacy of ibrutinib for the treatment of AIHA in adult patients with CLL/SLL or CLL-like MBL.

Patients will receive ibrutinib 420 mg/day PO for up to 12 cycles of 28 days in the absence of CLL progression or unacceptable toxicity. Every patient will be followed-up for 1 year after the completion of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CLL/small lymphocytic lymphoma (SLL) or CLL-like monoclonal B-cell lymphocytosis (MBL) according to IWCLL guidelines.
2. Patients >18 years old
3. Active AIHA (wAIHA or CAD) that i) is relapsed after previous treatment with corticosteroids (with or without rituximab), or ii) is steroid-resistant (failure to obtain hematologic response within 3 weeks on at least 1 mg/kg predniso(lo)ne), or iii) is steroid-dependent (need to continue on predniso(lo)ne at a dose of >10 mg/day to maintain a response). AIHA is defined as: anemia (hemoglobin ≤10 g/dL; or hemoglobin >10 g/dL dependent on transfusions to maintain this level of hemoglobin) and laboratory evidence of hemolysis (presence of 3 of 4 markers: increased reticulocyte count, increased indirect bilirubin, increased lactate dehydrogenase, decreased haptoglobin) and positive DAT (either IgG DAT, C3 DAT or both).
4. Eligibility of patients with DAT-negative active AIHA should be confirmed by the Principal Investigator and co-Principal Investigator for the trial.
5. Signed written informed consent according to ICH/EU/GCP and national local laws.

Exclusion Criteria:

1. Contraindication to ibrutinib therapy as per treating physician's discretion.
2. Contraindication to ibrutinib therapy as per ibrutinib data sheet (severe hepatic impairment, known allergy to the drug or to one of the excipients, concomitant treatment with warfarin or other vitamin K antagonists).
3. Previous exposure to ibrutinib as CLL-directed therapy.
4. Other CLL/SLL- or AIHA-directed treatment at the time of enrollment in the study, other than corticosteroids.
5. Female patients who are currently in pregnancy or are willing to be pregnant or are lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Ibrutinib efficacy in terms of Overall response rate | at month 6
  Evaluation of the efficacy of ibrutinib therapy for the treatment of AIHA in patients with CLL/SLL or CLL-like MBL in terms of percentage of patients who achieved response (CR + PR)

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Ematologia Osp Careggi, Florence
  - Ematologia Osp Maggiore della Carità, Novara
  - Ematologia Osp Molinette, Torino